CLINICAL TRIAL: NCT04447989
Title: Safety of Sildenafil in Premature Infants With Severe Bronchopulmonary Dysplasia
Acronym: SILDI-SAFE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Christoph Hornik (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Christoph Hornik, Associate Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00104901; 1R61HL147833-01 (NIH)
Record Dates: First submitted 2020-06-22; First posted 2020-06-25 (Actual); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Bronchopulmonary Dysplasia of Newborn
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: Premature infants with severe BPD (inpatient in neonatal intensive care units) will be randomized in a dose escalating approach 3:1 (sildenafil: placebo) sequentially, into each of 3 cohorts. There will be approximately 40 randomized and dosed participants in each cohort for a total of up to 120 participants.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study drug (sildenafil or placebo) will be prepared in the pharmacy by the unblinded pharmacist. Treatment cohort will be randomly assigned electronically and communicated to the pharmacist via the study portal. All other study staff and the patients/parents will be blinded to the treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1, sildenafil (Active Comparator): Sildenafil (0.5 mg/kg IV or 1 mg/kg enteral) every 8 hours for 28 days
  Interventions: Drug: Sildenafil
- Cohort 1, placebo (Placebo Comparator): Placebo (IV or enteral) every 8 hours for 28 days
  Interventions: Drug: Placebo
- Cohort 2, sildenafil (Active Comparator): Sildenafil (1 mg/kg IV or 2 mg/kg enteral) every 8 hours for 28 days
  Interventions: Drug: Sildenafil
- Cohort 2, placebo (Placebo Comparator): Placebo (IV or enteral) every 8 hours for 28 days
  Interventions: Drug: Placebo
- Cohort 3, sildenafil (Active Comparator): Sildenafil (2 mg/kg IV or 4 mg/kg enteral) every 8 hours for 28 days
  Interventions: Drug: Sildenafil
- Cohort 3, placebo (Placebo Comparator): Placebo (IV or enteral) every 8 hours for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil — Sildenafil citrate injection or powder for suspension
  Other Names: Revatio
  Arms: Cohort 1, sildenafil; Cohort 2, sildenafil; Cohort 3, sildenafil
Drug: Placebo — dextrose 5%
  Other Names: Dextrose 5%
  Arms: Cohort 1, placebo; Cohort 2, placebo; Cohort 3, placebo

SUMMARY:
This is a multicenter, randomized, placebo-controlled, sequential dose-escalating, double-masked, safety study of sildenafil in premature infants (inpatient in Neonatal Intensive Care Units (NICUs)) with severe bronchopulmonary dysplasia (BPD).

DETAILED DESCRIPTION:
Screening/Baseline

Research staff will document informed consent from the parent/guardian for all participants who satisfy eligibility criteria. The following information will be recorded in the case report form (eCRF) from the clinical medical record:

1. Participant demographics, including birth weight and gestational age at birth
2. Maternal race/ethnicity
3. Medical history
4. Physical examination, including actual weight
5. All mean arterial pressure (MAP) obtained in the 24 hours before the first dose
6. Concomitant medications (within 24 hours prior to start of study drug)
7. Respiratory assessment
8. Laboratory evaluations
9. Echocardiogram: If performed per local standard of care < 14 days prior to start of study drug, a study-specific echocardiogram need not be repeated. If not performed per local standard of care < 14 days prior to start of study drug, an echocardiogram will be required to confirm eligibility.
10. Cardiac catheterization reports, if performed per local standard of care < 14 days prior to start of study drug.
11. Adverse events following initial study-specific procedure

Treatment Period

The treatment period will include Days 1-28 or last day of study drug if early withdrawal of study drug. The following information will be collected and recorded while the participant is on study drug:

1. Actual weight on study Days 7 (± 1 day), 14 (± 1 day), 21 (± 1 day), and 28 (± 1 day) of study drug administration
2. Date, time, amount, and route of study drug dose
3. All concomitant medications
4. MAP

   A. All MAP values obtained 24 hours after the first dose of study drug regardless of administration route.

   B. MAP values will be obtained at a minimum at the following time points i. Prior to the first dose of study drug or dose escalation: 2 hours (± 5 minutes), 1 hour (± 5 minutes), and 15 minutes (± 5 minutes) ii. If administration route is IV:
   1. During and following the first dose of study drug or dose escalation: MAP at start of infusion, every 15 minutes (± 5 minutes) during infusion, at end of infusion (inclusive of flush) (± 5 minutes), at 15 and 30 minutes (± 5 minutes) after end of infusion, hourly (± 15 minutes) for 4 hours, and once in the remaining 2 hours prior to the next dose.
   2. For subsequent IV doses, the lowest valid MAP value should be recorded daily while on study drug.

   iii. If the administration route is enteral:
   1. During and following the first dose of study drug or dose escalation: MAP at start of enteral administration, then every 15 minutes (± 5 minutes) for 90 minutes (1.5 hours), then every 30 minutes (± 5 minutes) for 60 minutes (1 hour), then hourly (± 15 minutes) for 4 hours, then once in the remaining 2 hours prior to the next dose.
   2. For subsequent enteral doses, the lowest valid MAP value should be recorded daily while on study drug.
5. Respiratory assessment, weekly
6. Laboratory evaluations, at least every other week
7. Echocardiograms and cardiac catheterization reports, if performed per local standard of care
8. Pharmacokinetic (PK) sampling (after Day 7)
9. Adverse events

Weaning Period (Cohorts 2 and 3)

The weaning period will begin following Day 28 of study drug or, following the last day of study drug if participant was withdrawn from study drug prior to Day 28 and the dose escalated to ≥ 0.5 mg/kg IV or ≥ 1 mg/kg enteral.

The following information will be collected and recorded while the participant is weaning from study drug:

1. Date, time, amount and route of study drug dose
2. MAP (the lowest MAP value on last day of wean should be recorded).
3. Respiratory assessment on last day of wean
4. Echocardiogram and cardiac catheterization reports, if performed per local standard of care
5. Adverse events

Follow-up Period

The follow-up period will include Days 1-28 after the last study drug dose; last study drug dose may occur prior to Day 28 for those participants who withdraw from study drug early; on Day 28 for those participants who complete the full treatment period; or after last weaning dose for those participants who require weaning. The following information will be reported in electronic data capture system (EDC) at Day 1 (+ 2 days) and 14 (± 2days) of the follow-up period (or days closest to and after Day 1 and 14, if >1 assessment is available), except for MAP, adverse events (AEs), and serious adverse events (SAEs) (which will be reported from Days 1-28 post last study drug dose) and standard of care echocardiograms or cardiac catheterization reports:

1. Physical examination, including actual weight
2. MAP (the lowest valid MAP value on follow-up Day 1, 14, 21, and 28 should be recorded).
3. Respiratory assessment
4. Laboratory evaluations
5. Echocardiogram on follow-up Day 1 (+2 days). If performed per local standard of care, a study-specific echocardiogram need not be repeated. If not performed per local standard of care on Day 1 (+2 days) of the follow-up period, an echocardiogram will need to be performed.
6. Echocardiograms and cardiac catheterization reports, if performed per local standard of care (during follow-up Days 1-28)
7. Adverse events and SAEs (during follow-up Days 1-28)

Final Study Assessment

Final study assessment will occur at the time of discharge or transfer. The following information will be collected:

1. Physical examination, including actual weight
2. Respiratory assessment
3. Echocardiogram and cardiac catheterization reports, if performed per local standard of care on the day of discharge or transfer or up to 2 days prior.
4. Global rank
5. Discharge information A. Discharge or transfer B. Death C. Duration of hospitalization
6. Record if treatment for retinopathy of prematurity (ROP) was required

ELIGIBILITY:
Inclusion Criteria:

1. Documented informed consent from parent or guardian, prior to study procedures
2. < 29 weeks gestational age at birth
3. 32-44 weeks postmenstrual age
4. Receiving respiratory support at enrollment:

   * If 32 0/7-35 6/7 weeks postmenstrual age: mechanical ventilation (high frequency or conventional)
   * If 36 0/7-44 6/7 weeks postmenstrual age: mechanical ventilation (high frequency or conventional) OR continuous positive airway pressure (CPAP)

Note:

* Criteria 3 and 4 define severe BPD for the purposes of this study
* CPAP is defined as any of the following:

  * Nasal cannula > 2 liters per minute (LPM)
  * Nasal continuous positive airway pressure (NCPAP)
  * Nasal intermittent positive pressure ventilation (NIPPV)
  * Noninvasive neurally adjusted ventilatory assist (NAVA)
  * Any other device designed to provide positive pressure through a nasal device (e.g., RAM cannula, etc.)

Exclusion Criteria:

1. Previous enrollment and dosing in this study, protocol number (NHLBI-2019-SIL), "Safety of Sildenafil in Premature Infants with Severe Bronchopulmonary Dysplasia (BPD)"
2. Previous exposure to sildenafil within 7 days prior to randomization*
3. Previous exposure to vasopressors within 24 hours prior to randomization*
4. Previous exposure to inhaled nitric oxide within 24 hours prior to randomization*
5. Previous exposure to milrinone within 24 hours prior to randomization*
6. Evidence of pulmonary hypertension or moderate/large patent ductus arteriosus (PDA) on the most recent echocardiogram performed within 14 days prior to randomization
7. Known major congenital heart defect requiring medical or surgical intervention in the neonatal period
8. Known allergy to sildenafil
9. Known sickle cell disease
10. Aspartate aminotransferase (AST) > 225 U/L < 72 hours prior to randomization
11. Alanine aminotransferase (ALT) > 150 U/L < 72 hours prior to randomization
12. Any condition that would make the participant, in the opinion of the investigator, unsuitable for the study.

    * Participant will be reassessed prior to dosing to reconfirm eligibility criteria.

Max Age: 29 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 125 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2025-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Hornik, MD, Principal Investigator — Duke UMC; Matt Laughon, MD, Principal Investigator — UNC
Locations (25):
- United States (25):
  - Arkansas Children's Research Institute, Little Rock, Arkansas
  - University of Arkansas Medical Sciences, Little Rock, Arkansas
  - Rady Children's Hospital and Health Center, San Diego, California
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - University of Florida Jacksonville Shands Medical Center, Jacksonville, Florida
  - Wolfson Children's Hospital, Jacksonville, Florida
  - Emory Children's Center, Atlanta, Georgia
  - Lurie Children's Hospital, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - University of Louisville School of Medicine, Louisville, Kentucky
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Childrens Mercy Hospital, Kansas City, Missouri
  - Children's Hospital of Nevada at University Medical Center, Las Vegas, Nevada
  - University of Rochester School of Medicine Children's Hospital, Rochester, New York
  - Westchester Medical Center - New York Medical College, Valhalla, New York
  - University of NC at Chapel Hill, Chapel Hill, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - University of Texas Health, Austin, Texas
  - Women's Hospital of Texas, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers

REFERENCES:
- [Background] Gonzalez D, Laughon MM, Smith PB, Ge S, Ambalavanan N, Atz A, Sokol GM, Hornik CD, Stewart D, Mundakel G, Poindexter BB, Gaedigk R, Mills M, Cohen-Wolkowiez M, Martz K, Hornik CP; Best Pharmaceuticals for Children Act - Pediatric Trials Network Steering Committee. Population pharmacokinetics of sildenafil in extremely premature infants. Br J Clin Pharmacol. 2019 Dec;85(12):2824-2837. doi: 10.1111/bcp.14111. Epub 2019 Dec 15. PMID 31475367
- [Background] Stoll BJ, Hansen NI, Bell EF, Walsh MC, Carlo WA, Shankaran S, Laptook AR, Sanchez PJ, Van Meurs KP, Wyckoff M, Das A, Hale EC, Ball MB, Newman NS, Schibler K, Poindexter BB, Kennedy KA, Cotten CM, Watterberg KL, D'Angio CT, DeMauro SB, Truog WE, Devaskar U, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Trends in Care Practices, Morbidity, and Mortality of Extremely Preterm Neonates, 1993-2012. JAMA. 2015 Sep 8;314(10):1039-51. doi: 10.1001/jama.2015.10244. PMID 26348753
- [Background] Jobe AH, Bancalari E. Bronchopulmonary dysplasia. Am J Respir Crit Care Med. 2001 Jun;163(7):1723-9. doi: 10.1164/ajrccm.163.7.2011060. No abstract available. PMID 11401896
- [Background] Khemani E, McElhinney DB, Rhein L, Andrade O, Lacro RV, Thomas KC, Mullen MP. Pulmonary artery hypertension in formerly premature infants with bronchopulmonary dysplasia: clinical features and outcomes in the surfactant era. Pediatrics. 2007 Dec;120(6):1260-9. doi: 10.1542/peds.2007-0971. PMID 18055675
- [Background] Morrow CB, McGrath-Morrow SA, Collaco JM. Predictors of length of stay for initial hospitalization in infants with bronchopulmonary dysplasia. J Perinatol. 2018 Sep;38(9):1258-1265. doi: 10.1038/s41372-018-0142-7. Epub 2018 Jun 8. PMID 29880793
- [Background] Jackson W, Hornik CP, Messina JA, Guglielmo K, Watwe A, Delancy G, Valdez A, MacArthur T, Peter-Wohl S, Smith PB, Tolia VN, Laughon MM. In-hospital outcomes of premature infants with severe bronchopulmonary dysplasia. J Perinatol. 2017 Jul;37(7):853-856. doi: 10.1038/jp.2017.49. Epub 2017 Apr 6. PMID 28383537
- [Background] Poets CF, Lorenz L. Prevention of bronchopulmonary dysplasia in extremely low gestational age neonates: current evidence. Arch Dis Child Fetal Neonatal Ed. 2018 May;103(3):F285-F291. doi: 10.1136/archdischild-2017-314264. Epub 2018 Jan 23. PMID 29363502
- [Background] Tyson JE, Wright LL, Oh W, Kennedy KA, Mele L, Ehrenkranz RA, Stoll BJ, Lemons JA, Stevenson DK, Bauer CR, Korones SB, Fanaroff AA. Vitamin A supplementation for extremely-low-birth-weight infants. National Institute of Child Health and Human Development Neonatal Research Network. N Engl J Med. 1999 Jun 24;340(25):1962-8. doi: 10.1056/NEJM199906243402505. PMID 10379020
- [Background] Schmidt B, Roberts RS, Davis P, Doyle LW, Barrington KJ, Ohlsson A, Solimano A, Tin W; Caffeine for Apnea of Prematurity Trial Group. Caffeine therapy for apnea of prematurity. N Engl J Med. 2006 May 18;354(20):2112-21. doi: 10.1056/NEJMoa054065. PMID 16707748
- [Background] Doyle LW, Ehrenkranz RA, Halliday HL. Early (< 8 days) postnatal corticosteroids for preventing chronic lung disease in preterm infants. Cochrane Database Syst Rev. 2014 May 13;(5):CD001146. doi: 10.1002/14651858.CD001146.pub4. PMID 24825456
- [Derived] Schneider S, Bailey M, Spears T, Esther CR Jr, Laughon MM, Hornik CP, Jackson W. Safety of sildenafil in premature infants with severe bronchopulmonary dysplasia (SILDI-SAFE): a multicenter, randomized, placebo-controlled, sequential dose-escalating, double-masked, safety study. BMC Pediatr. 2020 Dec 14;20(1):559. doi: 10.1186/s12887-020-02453-7. PMID 33317479

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1, Sildenafil: Sildenafil was administered every eight hours in the following doses: 0.25 mg/kg IV or 0.5 mg/kg enteral on study days 1-2, 0.5 mg/kg IV or 1 mg/kg enteral on study days 3-28.
- Cohort 2, Sildenafil: Sildenafil was administered every eight hours in the following doses: 0.25 mg/kg IV or 0.5 mg/kg enteral on study days 1-2, 0.5 mg/kg IV or 1 mg/kg enteral on study days 3-4, 0.75 mg/kg IV or 1.5 mg/kg enteral on study days 5-6, 1 mg/kg IV or 2 mg/kg enteral on study days 7-28.
  A weaning schedule was used following the last study dose on Day 28 or if the patient was withdrawn from the study and escalated to a dose > 0.5 mg/kg IV or 1 mg/kg enteral. Whether IV or enteral, the weaning schedule was 75% of the last study dose on weaning days 1-2, 50% of the last study dose on weaning days 3-4, 25% of the last study dose on weaning days 5-6, and the weaning schedule was discontinued on weaning day 7.
- Cohort 3, Sildenafil: Sildenafil was administered every eight hours in the following doses: 0.25 mg/kg IV or 0.5 mg/kg enteral on study days 1-2, 0.5 mg/kg IV or 1 mg/kg enteral on study days 3-4, 0.75 mg/kg IV or 1.5 mg/kg enteral on study days 5-6, 1 mg/kg IV or 2 mg/kg enteral on study days 7-8, 1.25 mg/kg IV or 2.5 mg/kg enteral on study days 9-10, 1.5 mg/kg IV or 3 mg/kg enteral on study days 11-12, 1.75 mg/kg IV or 3.5 mg/kg enteral on study days 13-14, 2 mg/kg IV or 4 mg/kg enteral on study days 15-28.
  A weaning schedule was used following the last study dose on Day 28 or if the patient was withdrawn from the study and escalated to a dose > 0.5 mg/kg IV or 1 mg/kg enteral. Whether IV or enteral, the weaning schedule was 75% of the last study dose on weaning days 1-2, 50% of the last study dose on weaning days 3-4, 25% of the last study dose on weaning days 5-6, and the weaning schedule was discontinued on weaning day 7.
- Placebo: Placebo (IV or enteral) every 8 hours for 28 days
  Placebo: dextrose 5%
Period: Overall Study
Arm/Group | Cohort 1, Sildenafil | Cohort 2, Sildenafil | Cohort 3, Sildenafil | Placebo
Started | 32 | 30 | 32 | 31
Completed | 31 | 27 | 31 | 26
Not Completed | 1 | 3 | 1 | 5
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Transfer | 0 | 1 | 0 | 0
Not completed — Discharge | 0 | 1 | 1 | 3
Not completed — Ineligibility | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) population
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1, Sildenafil | Cohort 2, Sildenafil | Cohort 3, Sildenafil | Placebo | Total
Number analyzed (Participants) | 32 | 29 | 32 | 31 | 124
Age, Customized [Mean (Standard Deviation); unit: weeks]
  Gestational age | 25.16 (1.46) | 25.49 (1.70) | 25.40 (1.59) | 25.45 (1.76) | 25.37 (1.61)
  Postnatal age | 13.21 (3.44) | 12.44 (3.12) | 11.96 (3.54) | 12.48 (3.43) | 12.53 (3.38)
  Post-menstrual age | 38.37 (2.84) | 37.94 (3.19) | 37.37 (2.73) | 37.94 (3.27) | 37.90 (3.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 16 | 9 | 59
  Male | 15 | 12 | 16 | 22 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2 | 1 | 5
  Not Hispanic or Latino | 28 | 28 | 27 | 27 | 110
  Unknown or Not Reported | 2 | 1 | 3 | 3 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 29 | 32 | 31 | 124

OUTCOME MEASURES:

1. Primary Outcome: Safety Based Upon Number of Participants With Hypotension
Description: Safety as determined by incidence of hypotension experienced by the participants through 28 days post last dose of study drug.
  Hypotension will be defined as any clinically significant low blood pressure event deemed by the treating physician to require intervention with a fluid bolus or the initiation or escalation of inotropic, vasopressor, or systemic steroid therapy with the specific intent to raise blood pressure.
Time Frame: 28 days post last dose of study drug, up to 9 weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Sildenafil | Cohort 2, Sildenafil | Cohort 3, Sildenafil | Placebo
Number analyzed (Participants) | 31 | 29 | 32 | 30
Participants | 1 | 0 | 0 | 0

2. Secondary Outcome: Central Volume of Distribution (Vc) Population Pharmacokinetics (popPK)
Time Frame: Following the completion of 7 days (168 hours) of study drug administration
Population: Population Pharmacokinetics (popPK) analysis does not involve separating PK parameters by dose group. All samples across all dose groups are analyzed together.
Measure: Median (95% Confidence Interval); unit: L
Groups:
- Pharmacokinetics (PK) Cohort: Infants with samples collected who received at least one dose of sildenafil.
Arm/Group | Pharmacokinetics (PK) Cohort
Number analyzed (Participants) | 85
L | 3.86 [1.28 to 11.07]

3. Secondary Outcome: Peripheral Volume of Distribution (Vp) Population Pharmacokinetics (popPK)
Time Frame: Following the completion of 7 days (168 hours) of study drug administration
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: L
Arm/Group | Pharmacokinetics (PK) Cohort
Number analyzed (Participants) | 85
L | 4.49 [2.87 to 6.66]

4. Secondary Outcome: Clearance Population Pharmacokinetics (popPK)
Time Frame: Following the completion of 7 days (168 hours) of study drug administration
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: L/h
Arm/Group | Pharmacokinetics (PK) Cohort
Number analyzed (Participants) | 85
L/h | 2.69 [1.00 to 7.94]

5. Secondary Outcome: Half-life Population Pharmacokinetics (popPK)
Time Frame: Following the completion of 7 days (168 hours) of study drug administration
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Pharmacokinetics (PK) Cohort
Number analyzed (Participants) | 85
hours | 8.79 [8.00 to 9.42]

6. Secondary Outcome: Peak Plasma Concentration Population Pharmacokinetics (popPK)
Time Frame: Following the completion of 7 days (168 hours) of study drug administration
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Pharmacokinetics (PK) Cohort
Number analyzed (Participants) | 85
ng/mL | 130.5 [70.9 to 256.0]

7. Other Pre Specified Outcome: Number of Participants at Each Global Rank
Description: Global rank is defined as clinically significant events ranked in order of decreasing perceived severity. Rank descriptions are presented from most to least severe.
Time Frame: 28 days post last dose of study drug, up to 9 weeks
Population: Intent to treat (ITT) population with a global rank available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, Sildenafil | Cohort 2, Sildenafil | Cohort 3, Sildenafil | Placebo
Number analyzed (Participants) | 31 | 29 | 32 | 30
Participants
  Mortality | 0 | 2 | 1 | 0
  Extracorporeal life support | 0 | 0 | 0 | 0
  Tracheostomy | 8 | 3 | 4 | 9
  Periventricular leukomalacia (PVL) | 1 | 1 | 0 | 0
  Seizures | 1 | 2 | 1 | 1
  Dialysis | 0 | 0 | 0 | 0
  Retinopathy of prematurity (ROP) | 13 | 11 | 18 | 12
  Short gut syndrome/intestinal failure | 0 | 0 | 0 | 0
  Ventriculoperitoneal (VP) shunt | 0 | 0 | 0 | 0
  Gastrostomy tube | 4 | 2 | 3 | 1
  Surgical necrotizing enterocolitis/intestinal perforation (NEC/IP) | 0 | 0 | 0 | 0
  Patent ductus arteriosus (PDA) | 0 | 1 | 2 | 2
  Meningitis | 0 | 0 | 0 | 0
  Sepsis | 0 | 1 | 0 | 0
  Duration of hospitalization >= 52 weeks PMA | 0 | 0 | 0 | 0
  Duration of hospitalization 48 - 51 weeks PMA | 1 | 3 | 0 | 0
  Duration of hospitalization 44 - 47 weeks PMA | 1 | 2 | 1 | 2
  Duration of hospitalization 40 - 43 weeks PMA | 2 | 1 | 2 | 2
  Duration of hospitalization 36 - 39 weeks PMA | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 28 days post last dose of study drug, up to 9 weeks
Description: Serious Adverse Events were collected on the safety population. Non-serious Adverse Events were not collected per protocol.
Arm/Group | Cohort 1, Sildenafil | Cohort 2, Sildenafil | Cohort 3, Sildenafil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 2/29 | 1/32 | 0/30
Serious Adverse Events (participants affected / at risk) | 3/31 | 0/29 | 4/32 | 4/30
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1, Sildenafil (N=31) | Cohort 2, Sildenafil (N=29) | Cohort 3, Sildenafil (N=32) | Placebo (N=30)
Retinopathy of prematurity (Eye disorders) | 2 | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Meningitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Streptococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Cardiac dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Weaning failure (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/89/NCT04447989/Prot_SAP_001.pdf
  • Informed Consent Form (2024-03-27): https://cdn.clinicaltrials.gov/large-docs/89/NCT04447989/ICF_000.pdf